CLINICAL TRIAL: NCT05764447
Title: Improving Chemotherapy-induced Peripheral Neuropathy in Cancer Patients Using a Combined Qigong Baduanjin and Self-administered Acupressure Intervention: A Randomized Controlled Trial
Brief Title: Combined Qigong and Acupressure for Improving Chemotherapy-induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Shuk-Ting, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW22587
Record Dates: First submitted 2023-02-14; First posted 2023-03-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: cancer; neuropathy; acupressure; qigong; Baduanjin; chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent randomizer will prepare a computer-generated list of random assignments in sealed, sequentially numbered opaque envelopes. To aid allocation concealment, permuted blocks of varying sizes with an allocation weight of 1:1 will be used. The randomizer will keep a secure copy of the randomization list, which will be concealed from all research personnel and participants. The statistician performing data analysis will be blinded. Although it is not feasible to blind the participants or intervention personnel to the group assignments, the outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Qigong Baduanjin and Self-administered Acupressure Intervention (Experimental): The intervention will last 16 weeks, including twice-weekly supervised group sessions. The first 8 weeks will focus on training of qigong Baduanjin and self-administered acupressure. The duration of each group session will be 90 min. From week 9 onwards, the group sessions will be shortened to 60 min twice a week led by the BQ master. For self-practice prescription, participants will be instructed to practice the combined BQ and acupressure intervention three times a week (30 min each time) on the days without group sessions.
  Interventions: Behavioral: Combined qigong Baduanjin and self-administered acupressure
- Wait-list Control Group (Active Comparator): The control group will be offered a free modality of their choice after the last follow-up. The participants will receive usual care alone during the study period.
  Interventions: Behavioral: Wait-list Control

INTERVENTIONS:
Behavioral: Combined qigong Baduanjin and self-administered acupressure — The intervention will combine Baduanjin (BQ) and acupressure. The general design of the combination intervention is for BQ to be performed first (20 min), followed by self-administered acupressure (10 min). BQ comprises eight simple standardized movements. The combination of these simple body movements, breath control, and mindful meditation is designed to improve qi function.The acupressure protocol comprises six acupoints, i.e., Hegu, Quchi, Zusanli, Sanyinjiao, Qihai, and Taichong, which are the most commonly used acupoints in acupuncture trials for relieving CIPN according to previous reviews. These acupoints, based on TCM theory, are beneficial for strengthening the origin of qi and directing its flow to the upper and lower extremities. A massage pen will be used to stimulate the acupoints because participants with CIPN may have difficulty applying pressure with their hands/fingers.
  Arms: Combined Qigong Baduanjin and Self-administered Acupressure Intervention
Behavioral: Wait-list Control — The participants will receive usual care alone during the study period and will be offered the training after the last follow-up.
  Arms: Wait-list Control Group

SUMMARY:
The objective of the study is to investigate the effects of a 16-week combined qigong and acupressure intervention on reducing self-reported chemotherapy-induced peripheral neuropathy (CIPN) severity, objective measures of CIPN severity, lower-extremity functioning, handgrip strength, fall incidence, and health-related quality of life post-intervention among post-chemotherapy adult cancer patients. This will be a 2-arm assessor-blinded randomized controlled trial that will follow the CONSORT guidelines. A total of 104 cancer patients aged ≥18 who have completed neurotoxic chemotherapy at least 1 month prior to enrolment and experiencing CIPN will be recruited and randomized into combined qigong and self-administered acupressure intervention and wait-list control groups. The intervention group comprises of twice-weekly supervised group sessions and three times-weekly self-practice prescription (30 min each time) on days without group sessions. The control group will be offered a free modality of their choice after the last follow-up. The participants will receive usual care alone during the study period.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most common side effects of chemotherapy experiencing by cancer patients. CIPN can lead to significant distress, diminished health-related quality of life, functional decline, and an increased risk of falls in cancer patients, as they may experience altered proprioception. CIPN may continue to progress for several months post-treatment or even persist for years following chemotherapy.

Current pharmacological approaches are limited not only by side effects (e.g., fatigue, dizziness, insomnia, or nausea) but also by patients' unwillingness to further medicate a drug-related side effect. Also, the drugs may treat pain but not non-painful CIPN symptoms, and cannot induce neuro-protection or neuro-regeneration. Non-pharmacological interventions may be more appealing to patients, as they usually have no side effects and may result in clinical benefits for CIPN sufferers.

Acupressure is a non-invasive variant of acupuncture both adopting the meridian theory of traditional Chinese medicine (TCM) that stimulate acupoints across meridians and facilitate the flow of qi (energy) and blood, thereby restoring health and treating disease. Qigong is a mind-body exercise also rooted in the meridian theory of TCM. Through a combination of movement, breath control, and meditation, meridians can be opened, and the flow of qi and blood stimulated, to restore health. The combination approach is likely to elicit complementary physiologic adaptations on mechanisms involving both the peripheral and central nervous systems, thereby inducing a larger and potentially clinically meaningful improvement on CIPN.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* diagnosis of cancer
* completed neurotoxic chemotherapy at least 1 month prior to enrolment
* experiencing CIPN (defined as tingling, numbness, or pain in the extremities in the past week, on the basis of a score ≥4 on an 11-point numerical rating scale due to receiving neurotoxic chemotherapy)
* Eastern Cooperative Oncology Group performance status between 0 and 2
* able to communicate in Cantonese or Mandarin

Exclusion Criteria:

* they have psychiatric disorders or conditions that preclude practicing qigong or acupressure (e.g., recent myocardial infarction, breathing difficulties requiring oxygen use or hospitalization, cannot walk independently)
* have regularly engaged in qigong or acupressure (>once per week) in the previous 6 months
* are receiving acupuncture
* are pregnant or lactating
* have any infection/injury/ulcers around the acupoints, or had peripheral neuropathy before chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported CIPN severity post-intervention | Change from baseline (week 0) to post-intervention (week 16)
  The 11-item version of Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG Ntx) subscale will be used. It covers four domains: sensory, motor, hearing, and dysfunction. Items are rated on a scale of 0 (not at all) to 4 (very much), with higher scores indicating more severe CIPN. The Chinese version of FACT/GOG-Ntx has demonstrated satisfactory reliability and validity.

SECONDARY OUTCOMES:
Change in self-reported CIPN severity at follow-up | Change from baseline to 12 weeks after the intervention ends (week 28)
  The 11-item version of Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG Ntx) subscale will be used. It covers four domains: sensory, motor, hearing, and dysfunction. Items are rated on a scale of 0 (not at all) to 4 (very much), with higher scores indicating more severe CIPN. The Chinese version of FACT/GOG-Ntx has demonstrated satisfactory reliability and validity.
Objective CIPN severity | Change from baseline (week 0) to post-intervention (week 16), Change from baseline to 12 weeks after the intervention ends (week 28)
  The sensory nerve action potential amplitude (SNAP) and sensory nerve conduction velocity (SNCV) will be measured to reflect the objective CIPN severity using Mediracer Device, a hand-held device comprising stimulation electrodes, cables and analysis software. It has been validated for assessing carpel tunnel syndrome and used to quantify CIPN severity. The electrodes are attached to the wrist and the base of index finger. This device causes minimal discomfort to patients and can be used by trained research assistants. The lower SNAP and SNCV, the more severe CIPN.
Handgrip strength | Change from baseline (week 0) to post-intervention (week 16), Change from baseline to 12 weeks after the intervention ends (week 28)
  Handgrip strength will be measured by a dynamometer. The maximum reading of two trials in standing position with full elbow extension using the dominant hand will be taken
Lower-extremity physical functioning | Change from baseline (week 0) to post-intervention (week 16), Change from baseline to 12 weeks after the intervention ends (week 28)
  The Short Physical Performance Battery (SPPB) is an objective assessment tool used to measure lower-extremity physical functioning and is highly predictive of fall risk (44). It consists of 3 functional tasks which can be completed within 10 minutes. A summary score ranges from 0 to 12, with a higher score indicating a higher level of physical functioning.
Fall incidence | post-intervention (week 16), 12 weeks after the intervention ends (week 28)
  Fall incidence will be assessed by patient self-reports. A fall is deﬁned as unintentionally coming to rest on the ground or at some other lower level. Participants indicating a fall will be asked about any resultant injury (e.g., sprains, fractures, head injuries) and the need to seek medical care.
Global health-related quality of life (HRQoL) | Change from baseline (week 0) to post-intervention (week 16), Change from baseline to 12 weeks after the intervention ends (week 28)
  Global HRQoL will be measured using the 27-item Functional Assessment of Cancer Therapy-General (FACT-G). It consists of 4 subscales: physical, emotional, social/family, and functional well-being. Each item is rated from 0 ("not at all") to 4 ("very much"). Higher score represent better HRQoL. FACT-G has been validated in Chinese populations with good reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request as decided by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 3 years after the manuscript on main findings is published.